CLINICAL TRIAL: NCT05191784
Title: A Phase 2, Open-label, Single-arm Study to Evaluate the Efficacy and Safety of GX-I7 in Combination With Bevacizumab in Recurrent Glioblastoma (GBM) Patients
Brief Title: GX-I7 in Combination With Bevacizumab in Recurrent Glioblastoma (GBM) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GX-I7-CA-010
Record Dates: First submitted 2021-11-10; First posted 2022-01-13 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — efineptakin alfa; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GX-I7 and bevacizumab (Experimental): Bevacizumab at a dose of 10 mg/kg intravenously, and GX-I7 intramuscularly.
  Interventions: Drug: GX-I7; Drug: Bevacizumab

INTERVENTIONS:
Drug: GX-I7 — Administered by intramuscular (IM) injection
  Other Names: rhIL-7-hyFc; Efineptakin alfa
Drug: Bevacizumab — Administered by intravenous (IV) injection
  Other Names: Avastin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of GX-I7 in combination with bevacizumab in subjects with recurrent glioblastoma.

DETAILED DESCRIPTION:
This is a phase 2 study designed to evaluate the efficacy and safety of GX-I7 in combination with bevacizumab in subjects with recurrent glioblastoma.

A total of 20 patients will be enrolled in the study and administered bevacizumab GX-I7. The study treatment will be continued for up to 6 cycles or until a progression of disease or unacceptable toxicity is confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years
2. Histologically diagnosed glioblastoma patients who have been confirmed the progression of disease after attempting standard therapy (RT/CCRT and/or adjuvant chemotherapy (TMZ))
3. Karnofsky Performance Status; KPS ≥ 60 or ECOG status 0-2
4. Life expectancy > 12 weeks
5. Adequate hematologic and end organ function

Exclusion Criteria:

1. Malignancies other than disease under study within 5 years prior to the first dose of study drug
2. Subjects who have received bevacizumab or other VEGF inhibitors prior to study participation
3. Body Mass Index (BMI) ≥ 30 kg/m2
4. Subjects confirmed intracranial hemorrhage with non-contrast CT or MRI
5. Clinically significant cardiovascular disease
6. History of arterial or venous thromboembolism 6 months prior to study participation
7. Uncontrolled hypertension (blood pressure ≥ 150/90 mmHg with appropriate antihypertensive therapy)
8. History of hypertensive crisis or hypertensive encephalopathy
9. Subjects receiving therapeutic anticoagulation (except low molecular weight heparin or warfarin)
10. Pregnancy or breastfeeding.
11. Subjects with active virus infection
12. Subjects with autoimmune disease/ syndromes
13. Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study
14. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
15. Severe infections during the screening period, including but not limited to complications of infection, bacteremia or severe pneumonia
16. Prior allogeneic bone marrow transplantation or prior solid organ transplantation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From the initiation of study treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Progression free survival (PFS) by iRANO criteria
Overall survival (OS) | From the initiation of study treatment until the date of death from any cause, assessed up to 24 months.
  Overall survival (OS)

SECONDARY OUTCOMES:
ORR (Objective response rate) | From the date of complete response or partial response until the date of first documented progression, assessed up to 24 months.
  ORR (Objective response rate) by iRANO criteria
DOR (Duration of response) | From the date of complete response or partial response until the date of first documented progression, assessed up to 24 months.
  DOR (Duration of response) by iRANO criteria
DCR (Disease control rate) | From the date of complete response, partial response, or stable disease until the date of first documented progression, assessed up to 24 months.
  DCR (Disease control rate) by iRANO criteria
Incidence of adverse events (AEs) | Through study completion, an average of 1 year
  The incidence rate of adverse events (AEs) graded according to NCI CTCAE v5.0
Immunogenicity (ADA) | Day 1 and Day 43 of each cycle (8-week interval)
  The incidence rate of anti-drug antibodies (ADAs)
Immunogenicity (neutralizing antibody) | Day 1 and Day 43 of each cycle (8-week interval)
  The incidence rate of anti-drug antibodies (neutralizing antibody)
Absolute counts and ratios of immune cell subtypes | Day 1 and Day 29 of each cycle (8-week interval)
  Changes of absolute counts and ratios of immune cell subtypes

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Heo, Study Director — Genexine, Inc.
Locations (1):
- Seoul St.Mary's Hospital of the Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No